CLINICAL TRIAL: NCT02226263
Title: Incidence of Severe Necrotizing Enterocolitis in Preterm Newborns <1500g Using Probiotics Lactobacillus Boucardii.
Brief Title: Severe Necrotizing Enterocolitis in Preterm Newborns <1500g Using Probiotics
Acronym: EPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Guadalupe Gómez Rodríguez, neonatologist, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: R-2010-1002-12
Record Dates: First submitted 2014-07-22; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Infectious Diseases
Keywords: Necrotizing enterocolitis; Probiotics; Preterm newborns
MeSH Terms: conditions — Communicable Diseases; Enterocolitis, Necrotizing | interventions — Biological Evolution; Drainage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- probiotics Lactobacillus acidophilus boucardii strain. (Experimental): Lactobacillus acidophilus boucardii strain was added at a dose of 125 mg/ kg/dose twice daily for 4 weeks .The probiotic presentation used was powder in an envelope with 160mg (Carnot ® Laboratories), scientific products, Mexico, (Registration Number 274M91SSA). This was stored in a dry place at room temperature, avoiding sunlight.
  Interventions: Dietary Supplement: probiotics Lactobacillus acidophilus boucardii

INTERVENTIONS:
Dietary Supplement: probiotics Lactobacillus acidophilus boucardii — Using sterile technique, the probiotic with 1x109 [CFU] Lactobacillus acidophilus boucardii strain was added at a dose of 125 mg/ kg/dose twice daily for 4 weeks to fresh supplement breast milk or formula for preterm infants.
  Other Names: Gastric tolerance, characteristics of discharges, evolution, reason for discharge, and the development of NEC was monitored.

SUMMARY:
The purpose of this study is to know the effects of probiotics on the incidence of Necrotizing Enterocolitis (NEC) in preterm infants less than 1500 g.

DETAILED DESCRIPTION:
The investigators performed a clinical, randomized, double-blind trial in preterm infants <1500g from March 1, 2010 to February 28, 2012. Group A received enteral stimulation trophic five days and later increments 20ml/k/day of breast milk or formula for premature; the group B apart from the above the probiotic Lactobacillus acidophilus (boucardii strain) 1 X109 colonic forming unit (CFU)/ day for 4 weeks was added. Gastric tolerance, evolution, reason for discharge, and the development of Necrotizing enterocolitis was monitored. The diagnosis of Necrotizing enterocolitis was made by the treating physician according to Bell's criteria and was blinded to group assignments.The formulas were prepared by one of the investigators according to the group each patient was assigned. Using sterile technique, the probiotic with 1x109 (CFU) Lactobacillus acidophilus (boucardii strain) was added at a dose of 125 mg/ kg/dose twice daily for 4 weeks to fresh supplement breast milk or formula for preterm infants. In case of control group only breast milk or formula for preterm infants was used.

All formulas were labeled for each patient and were delivered to the nurse in charge of infant feeding at 9:00 and 21:00 h.

Characteristics of Sample size and statistical analysis:

Sample size showed that the investigators needed 190 total preterm infants, based on the expected 50% decrease in the incidence of severe necrotizing enterocolitis in preterm neonates who received probiotics compared with control group with α 0.05 and β 0.20. Student´s t test or Mann Whitney U test were performed for mean differences regarding the general characteristics in the two study groups, Chi square or Fisher´s test for differences in proportions for mortality and complications between groups.

ELIGIBILITY:
Inclusion Criteria:

* We studied 150 preterm newborns <1500gr who were recruited on the day that began enteral feeding according to the decision of the treating physician.

Exclusion Criteria:

* Preterm infants > 1500g with Apgar score <6 at 5 minutes, gastrointestinal malformations, fetopathies, patent ductus arteriosis with hemodynamic decompensation, asphyxia, and NEC suspected as classified by Bell were excluded from the study.

Ages: 27 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2010-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Incidence of severe necrotizing enterocolitis in preterm newborns <1500g | 23 month
  Group A received enteral stimulation trophic five days and later increments 20ml/k/day of breast milk or formula for premature; the group B apart from the above the probiotic Lactobacillus boucardii 1 X109 (CFU) / day for 4 weeks was added.

SECONDARY OUTCOMES:
Adverse effects with probiotic use in preterm newborns <1500g. | 23 month
  The amount of food was increased slowly if tolerated according to the Clinical Practice Guidelines for enteral feeding preterm in our hospital, enteral feeding was interrupted if there was any sign of intolerance such as vomiting, presence of bile or blood content by probe orogastric, bloating, or bloody stools which were assessed and recorded daily.Our primary outcome was the presence of severe necrotizing enterocolitis (NEC) monitored by the Bell´s criteria; secondarily we evaluated the presence of sepsis diagnosed with clinical signs of systemic inflammatory response and positive blood culture.

OTHER OUTCOMES:
Diagnosis the Necrotizing Enterocolitis (NEC) | 23 month
  Our primary outcome was the presence of severe (NEC) monitored by the Bell´s criteria; secondarily we evaluated the presence of sepsis diagnosed with clinical signs of systemic inflammatory response and positive blood culture,

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Gómez, M.D., Principal Investigator — Universidad de Guanajuato
Locations (1):
- Instituto Mexicano del seguro social, León, Guanajuato, Mexico